CLINICAL TRIAL: NCT02032290
Title: Assessment of Coronary Flow Reserve by Doppler Flow Wire in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention Differences Between the Loading Dose of Ticagrelor and Clopidogrel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Massimo Mancone, PhD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Ticagrelor - Clopidogrel
Record Dates: First submitted 2013-12-18; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Acute Coronary Syndrome:; Non ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Angina, Unstable | interventions — Percutaneous Coronary Intervention

ARMS (2):
- ticagrelor (Active Comparator): ticagrelor: loading dose of 180 mg and maintaining dose of 90 mg twice daily in NSTEMI and STEMI (Class I B) patients;
  Interventions: Procedure: Assessment of Coronary Flow Reserve; Procedure: Percutaneous coronary intervention; Drug: ticagrelor loading
- clopidogrel (Active Comparator): clopidogrel: loading dose of 600 mg and maintaining dose of 75 mg daily in NSTEMI (Class I B) and STEMI (Class I C) patients.
  Interventions: Procedure: Assessment of Coronary Flow Reserve; Procedure: Percutaneous coronary intervention; Drug: Clopidogrel loading

INTERVENTIONS:
Procedure: Assessment of Coronary Flow Reserve
Procedure: Percutaneous coronary intervention
Drug: ticagrelor loading
  Arms: ticagrelor
Drug: Clopidogrel loading
  Arms: clopidogrel

SUMMARY:
The administration of these drugs is realized according to the European Society of Cardiology guidelines.

All patients will be pretreated with aspirin 300 mg orally, heparin iv to maintain an activated clotting time of >250 sec, and a loading dose of ticagrelor (180 mg) or clopidogrel (600 mg) immediately before the revascularization. The list of assignment to ticagrelor or clopidogrel will be generated by a computer according to a 1:1 randomization. Primary Percutaneous Coronary Intervention will be performed according to standard clinical practice using femoral or radial artery Judkins approach via six or seven French heath insertion. After crossing the target occlusive Lesion, coronary stenting will be performed based on standard practice. Patients subsequently will receive heparin for 48 hr, aspirin 100 mg daily, and clopidogrel (75 mg/day) or ticagrelor (90 mg twice daily) for at least 12 months. Other adjunctive pharmacotherapy in Intensive Care Unit will be administered according to operator discretion. All patients will provide written informed consent before entering the study.

Before and after the procedure a 12-leads ECG and an echocardiogram will be performed as standard practice. Then, all the pre-, intra-, and post-procedure data patients will be collected in a database.

Investigators aim to perform a prospective, single-center, investigator-initiated, randomized study to compare the Adenosine-induced coronary vasodilatation after the loading dose of Ticagrelor either Clopidogrel during the Percutaneous Coronary Intervention. Patients with Acute Coronary Syndrome undergoing Percutaneous Coronary Intervention will be enrolled in the study and will be randomized, in a 1:1 ratio, to receive a loading dose of Ticagrelor (180 mg) or Clopidogrel (600 mg). Coronary Flow Reserve will be recorded by intracoronary Doppler Flow Wire before the stent implantation and after the procedure at baseline and 2-minute later adenosine intravenous administration at incremental doses of 50, 80, 110 and 140 ug/Kg/min with 2 minutes interval between infusions.

Coronary Flow Reserve is the ability of the myocardium to increase blood flow in response to maximal exercise. Doppler Flow Wire allows to measure this increase expressing it as a ratio between maximal vasodilation and flow at rest. Coronary Flow Reserve is routinely measured in patients with Acute Coronary Syndrome, without an increased risk of adverse events for patients neither adjunctive costs for the National Health System.

Furthermore, Plasma concentrations of Ticagrelor and its main metabolite (AR-C124910XX) will be measured in venous blood collected at the end of the procedure. In patients requiring a second Percutaneous Coronary Intervention, for example for multivessel disease, all these measures will be repeated in the same manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndromes undergoing Percutaneous Coronary Intervention with stent implantation;
* Patients ≥ 18 and ≤ 75 years old.
* Signed informed consent;

Exclusion Criteria:

* Patients with stable angina;
* prior myocardial infarction;
* prior revascularization (Percutaneous Coronary Intervention or coronary artery bypass grafting);
* Clopidogrel and/or Ticagrelor contraindications (history of intracranial hemorrhage, active pathological bleeding, severe hepatic impairment);
* major periprocedural complications;
* Glomerular filtration rate < 30 ml/min or requiring haemodialysis;
* Non-sinus rhythm;
* severe chronic obstructive pulmonary disease;
* requirement for oral anticoagulant;
* risk of bleeding or bradycardic events;
* Ejection fraction < 45%;
* Cardiogenic shock;
* Severe left ventricular hypertrophy;
* severe valvular disease;
* indication to coronary artery bypass grafting;
* diffuse coronary atherosclerosis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
assessment of coronary flow reserve | 2 hours after the loading dose of drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Massimo Mancone, Rome, Rome, Italy